CLINICAL TRIAL: NCT03416894
Title: Deep Brain Stimulation (DBS) for the Treatment of Refractory Post-Traumatic Stress Disorder (PTSD): Pilot Trial
Brief Title: Deep Brain Stimulation for Treatment Refractory PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 165-2017
Record Dates: First submitted 2018-01-08; First posted 2018-01-31 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Brain Stimulation (Experimental)
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — DBS offers the opportunity to insert electrodes into deep brain structures and electrically stimulate them in a titratable and ultimately reversible manner

SUMMARY:
This is a phase I, non-blinded, non-randomized, pilot trial for safety and efficacy of deep brain stimulation for PTSD. A substantial number of individuals continue to experience PTSD symptoms despite appropriate medical treatment. In psychotherapy-based studies, over 30% of patients that completed a full course of treatment continue to meet criteria for PTSD. Response rates to treatment with SSRIs are usually no higher than 60%. This study would be the first exploration of a surgical therapy for refractory PTSD. The subgenual cingulate plays a role in mechanisms of this disorders and has been successfully targeted with DBS for the treatment of depression. The development of a therapy that targets brain structures known to play a role in this disease would be a substantial step forward in the treatment and understanding of these conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male patients between age 18-70
2. Diagnosis of posttraumatic stress disorder as defined by the Diagnostic and Statistical Manual fifth edition (DSM V).
3. Treatment Resistance as defined by the persistence of clinical symptoms despite adequate treatment with four modalities, including a) selective serotonin reuptake inhibitors, b) cognitive behavioral therapy, c) other classes of medications and/or psychotherapy.
4. Severe forms of the disease as measured by Clinician Administered PTSD scale (CAPS) scores ≥ 50.
5. A pattern of chronic stable PTSD lasting at least 1 year.
6. Ability to provide informed consent and comply with all testing, follow-ups and study appointments and protocols

Exclusion Criteria:

1. Any past or current evidence of psychosis or mania (patients with co-morbid depression will not be excluded from the study)
2. Active neurologic disease, such as epilepsy
3. Alcohol or substance dependence or abuse in the last 6 months, excluding caffeine and nicotine
4. Current suicidal ideation
5. Any contraindication to MRI or PET scanning
6. Likely to relocate or move out of the country during the study's one year duration
7. Presence of clinical and/or neurological conditions that may significantly increase the risk of the surgical procedure.
8. Currently pregnant (as determined by history and serum HCG) or lactating; for females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2018-01-19 (Actual); Primary Completion 2024-11-10 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events using SAFTEE collateral effects scale. | 1 year
  Adverse events (AE) will be recorded and categorized according to severity and relationship to procedure. All AEs will be assessed for their relationship to the study procedure.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD) | 1 year
  The HAMD is designed to rate the severity of depression in patients. 0-7 = Normal 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression
  ≥ 23 = Very Severe Depression
Beck's Depression Inventory (BDI) | 1 year
  BDI is a self-rated depression scale. 1-10:These ups and downs are considered normal;11-16: Mild mood disturbance; 17-20: Borderline clinical depression; 21-30: Moderate depression; 31-40: Severe depression; over 40: Extreme depression
Beck's Anxiety Inventory (BAI) | 1 year
  BAI is a self-rated anxiety scale. Score of 0 - 21 = low anxiety Score of 22 - 35 = moderate anxiety Score of 36 and above = potentially concerning levels of anxiety
Clinician-Administered PTSD Scale (CAPS) | 1 year
  The CAPS is a semi-structured interview that is designed to assess the essential features of Posttraumatic Stress Disorder.
Davidson Trauma Scale (DTS) | 1 year
  Self-report measure that assesses PTSD. The DTS yields a frequency score (ranging from 0 to 68), severity score (ranging from 0 to 68), and total score (ranging from 0 to 136). It can be used to make a preliminary determination about whether the symptoms meet DSM criteria for PTSD. Scores can also be calculated for each of the 3 PTSD symptom clusters (i.e., B, C, and D).
Short PTSD Rating Interview (SPRINT) | 1 year
  self-report measure that assesses the core symptoms of PTSD (intrusion, avoidance, numbing, arousal), somatic malaise, stress vulnerability, and role and social functional impairment. Symptoms are rates on five point scales from 0 (not at all) to 4 (very much).
Clinical Global Impression (CGI) | 1 year
  CGI is a 3-item observer-rated scale that measures illness severity (CGIS), global improvement or change (CGIC) and therapeutic response. The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). CGI-C scores range from 1 (very much improved) through to 7 (very much worse). Treatment response ratings should take account of both therapeutic efficacy and treatment-related adverse events and range from 0 (marked improvement and no side-effects) and 4 (unchanged or worse and side-effects outweigh the therapeutic effects). Each component of the CGI is rated separately; the instrument does not yield a global score.
Global Functioning Assessment (GFA) | 1 year
  GAF assigns a clinical judgment in numerical fashion to the individual's overall functioning level. Impairments in psychological, social and occupational/school functioning are considered, but those related to physical or environmental limitations are not.
  The scale ranges from 0 (inadequate information) to 100 (superior functioning).
36-Item Short Form Health Survey (SF-36) | 1 year
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting.
The State-Trait Anxiety Inventory (STAI) | 1 year
  STAI is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndrome. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Hamilton Anxiety Rating Scale (HAMA) | 1 year
  The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Sheehan disability scale (SDS) | 1 year
  The SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life. Total score 0-30 (0 unimpaired, 30 highly impaired) Work/school (0-10) Social life (0-10) Family life/home responsibilities (0-10 Scores of ≥5 on any of the 3 scales; high scores are associated with significant functional impairment.
Positive and negative affect (PANAS) | 1 year
  PANAS comprises two mood scales, one that measures positive affect and the other which measures negative affect. Used as a psychometric scale, the PANAS can show relations between positive and negative affect with personality stats and traits. Ten descriptors are used for each PA scale and NA to define their meanings.
  Participants in the PANAS are required to respond to a 20-item test using 5-point scale that ranges from very slightly or not at all (1) to extremely (5).

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No